CLINICAL TRIAL: NCT03678688
Title: A Phase 1/2, Active-controlled, Randomized, Open-label Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Multiple Oral Doses of OPC-167832 Tablets in Subjects With Uncomplicated, Smear-positive, Drug-susceptible Pulmonary Tuberculosis
Brief Title: A Phase 1/2 Trial of Multiple Oral Doses of OPC-167832 for Uncomplicated Pulmonary Tuberculosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 323-201-00003; OPP1178898 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary TB
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — OPC-67683

STUDY DESIGN:
Intervention Model Description: This will be a multiple-dose trial of OPC-167832 with 2 stages.
  Stage 1 is a multiple ascending dose trial planned to be conducted in 4 sequential cohorts of 18 participants each. There will be 2 arms (OPC-167832, combination of rifampicin, isoniazid, ethambutol, and pyrazinamide (RHEZ)) in each cohort.
  Stage 2 will be a parallel group comparison of 4 treatment regimens: 1) OPC-167832 plus Delamanid 2) OPC-167832 plus Bedaquiline 3) OPC-167832 plus Delamanid plus Bedaquiline 4) RHEZ.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Stage 1: RHEZ (Active Comparator): Participants received a single dose of RHEZ (each tablet containing 150 milligrams (mg) rifampicin, 75 mg isoniazid, 400 mg pyrazinamide, and 275 mg ethambutol), orally, once daily (QD) from Day 1 through Day 20.
  Interventions: Drug: RHEZ
- Stage 1: 10 mg OPC-167832 (Experimental): Participants received OPC-167832, 10 mg, orally, QD, from Day 1 through Day 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 10 mg OPC-167832
- Stage 1: 30 mg OPC-167832 (Experimental): Participants received OPC-167832, 30 mg, orally, QD from Day 1 through Day 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 30 mg OPC-167832
- Stage 1: 90 mg OPC-167832 (Experimental): Participants received OPC-167832, 90 mg, orally, QD from Day 1 through Day 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 90 mg OPC-167832
- Stage 1: 3 mg OPC-167832 (Experimental): Participants received OPC-167832, 3 mg, orally, QD from Day 1 through Day 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 3 mg OPC-167832
- Stage 2: 30 mg OPC-167832 + 300 mg Delamanid (Experimental): Participants received OPC-167832, 30 mg, in combination with delamanid, 300 mg, orally, QD from Day 1 through Day 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 30 mg OPC-167832 + 300 mg delamanid
- Stage 2: 30 mg OPC-167832 + 400 mg Bedaquiline (BDQ) (Experimental): Participants received OPC-167832, 30 mg, in combination with BDQ, orally, QD, from Day 1 through Day 14. Participants received a loading dose of 700 mg BDQ on Day 1 and 500 mg on Day 2. BDQ was then administered at a dose of 400 mg, QD, orally from Days 3 to 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 30 mg OPC-167832 + 400 mg BDQ
- Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ (Experimental): Participants received OPC-167832, 30 mg, in combination with delamanid, 300 mg and BDQ, 400 mg, orally, QD, from Day 1 through Day 14. Participants received a loading dose of 700 mg BDQ on Day 1 and 500 mg on Day 2. BDQ was then administered at a dose of 400 mg, orally, QD from Days 3 to 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
  Interventions: Drug: 30 mg OPC-167832 + 300 mg delamanid + 400 mg BDQ
- Stage 2: RHEZ (Active Comparator): Participants received a single dose of RHEZ (each tablet containing 150 mg rifampicin, 75 mg isoniazid, 400 mg pyrazinamide, and 275 mg ethambutol), orally, QD, from Day 1 through Day 20.
  Interventions: Drug: RHEZ

INTERVENTIONS:
Drug: 10 mg OPC-167832 — Once daily oral dose of 10 mg OPC-167832 from Day 1 through Day 14.
  Arms: Stage 1: 10 mg OPC-167832
Drug: 30 mg OPC-167832 — Once daily oral dose of 30 mg OPC-167832 from Day 1 through Day 14.
  Arms: Stage 1: 30 mg OPC-167832
Drug: 90 mg OPC-167832 — Once daily oral dose of 90 mg OPC-167832 from Day 1 through Day 14.
  Arms: Stage 1: 90 mg OPC-167832
Drug: 3 mg OPC-167832 — Once daily oral dose of 3 mg OPC-167832 from Day 1 through Day 14.
  Arms: Stage 1: 3 mg OPC-167832
Drug: RHEZ — RHEZ was used in both Stage 1 and Stage 2. Each tablet contains 150 mg rifampicin, 75 mg isoniazid, 400 mg pyrazinamide, and 275 mg ethambutol. Participants received a single-dose from Day 1 through Day 20. The total number of tablets per day was based on the pretreatment body weight:
  * Participants weighing 30 to 37 kg received 2 tablets per day
  * Participants weighing 38 to 54 kg received 3 tablets per day
  * Participants weighing 55 to 70 kg received 4 tablets per day
  * Participants weighing > 70 kg received 5 tablets per day
  Arms: Stage 1: RHEZ; Stage 2: RHEZ
Drug: 30 mg OPC-167832 + 300 mg delamanid — Once daily oral dose of 30 mg OPC-167832 plus 300 mg delamanid from Day 1 through Day 14.
  Arms: Stage 2: 30 mg OPC-167832 + 300 mg Delamanid
Drug: 30 mg OPC-167832 + 400 mg BDQ — Once daily oral dose of 30 mg OPC-167832 plus 400 mg BDQ from Day 1 through Day 14. Participants received a loading dose of 700 mg BDQ on Day 1 and 500 mg on Day 2. The dose of BDQ was 400 mg QD for Days 3 to 14.
  Arms: Stage 2: 30 mg OPC-167832 + 400 mg Bedaquiline (BDQ)
Drug: 30 mg OPC-167832 + 300 mg delamanid + 400 mg BDQ — Once daily oral dose of 30 mg OPC-167832 plus 300 mg delamanid plus 400 mg BDQ from Day 1 through Day 14. Participants received a loading dose of 700 mg BDQ on Day 1 and 500 mg on Day 2. The dose of BDQ was 400 mg QD for Days 3 to 14.
  Arms: Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ

SUMMARY:
This trial will evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of multiple oral doses of OPC-167832 in participants with uncomplicated, smear-positive, drug-susceptible pulmonary tuberculosis (TB).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written, informed consent prior to initiation of any trial-related procedures, and able, in the opinion of the investigator, to comply with all the requirements of the trial.
* Male or female participants between 18 and 64 years of age (inclusive) at the screening visit.
* Body mass index ≥ 16.0 and ≤ 32.0 kilograms per meters squared (kg/m^2) (inclusive) at the screening visit.
* Newly diagnosed, uncomplicated, drug-susceptible pulmonary TB.
* Microscopy performed on a sputum smear at screening indicates presence of acid-fast bacilli (at least 1+).
* Able to produce an adequate volume of sputum (approximately 10 millilitres (mL) or more estimated overnight production).
* Female participants of childbearing potential must agree to use 2 different approved methods of birth control or remain abstinent throughout the participation in the trial and for 12 weeks after the last dose of trial treatment (investigational medicinal product (IMP) or RHEZ).
* Male participants must agree to use 2 different approved methods of birth control or remain abstinent throughout the participation in the trial and for 12 weeks after the last dose of trial treatment (IMP or RHEZ).

Exclusion Criteria:

* Participants are known or suspected of having resistance to rifampicin, isoniazid, ethambutol, or pyrazinamide using any combination of Xpert Mycobacterium tuberculosis/Rifampin (MTB/RIF), line probe assay, culture, and/or epidemiologic history at screening.
* Poor general condition where no delay in treatment can be tolerated or where immediate hospital admission is warranted.
* Evidence of clinically significant metabolic (including ongoing or current hypokalemia), gastrointestinal, neurological, psychiatric, endocrine or liver (e.g., hepatitis B and C) disease; malignancy; or other abnormalities (other than the indication being studied).
* History of or current clinically relevant cardiovascular disorder such as heart failure, coronary heart disease, hypertension, arrhythmia or symptom strongly suggestive of such a problem (for example, syncope or palpitations), tachyarrhythmia or status after myocardial infarction.
* Known bleeding disorders or family history of bleeding disorders.
* Any diseases or conditions in which the use of delamanid, rifampicin, isoniazid, pyrazinamide, ethambutol, or Bedaquiline is contraindicated.
* Any prior treatment for M. tuberculosis within the past 3 years.
* Any treatment with a drug active against M. tuberculosis (e.g., quinolones) within the 3 months prior to screening.
* Clinical evidence of severe extrapulmonary TB (e.g., miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis).
* Evidence of pulmonary silicosis, lung fibrosis, or other lung condition considered as severe by the investigator (other than TB). In particular any underlying condition that could interfere with the assessment of x-ray images, sputum collection, or interpretation of sputum findings, or otherwise compromise the subject's participation in the trial.
* Any renal impairment characterized by serum creatinine clearance of <60 millilitres per minute (mL/min), or hepatic impairment characterized by alanine transaminase, aspartate transaminase, or total bilirubin >1.5 x upper limit of normal (ULN) of the clinical laboratory reference range at screening.
* For Stage 1, participants who are human immunodeficiency virus (HIV) positive are excluded. For Stage 2, participants with HIV co-infection who are on antiretroviral drugs during screening or with CD4 cell count <500/ millimeters cubed (mm^3) are excluded.
* Changes in the electrocardiogram (ECG) such as QTcF >450 milliseconds (msec), atrioventricular block II or III, bi-fasicular block, at screening or current history of clinically significant ventricular arrhythmias. Other ECG changes if considered clinically significant by the investigator.
* Participants receiving any of the prohibited medications within the specified periods or who would be likely to require prohibited concomitant therapy during the trial.
* Female participants who are breast-feeding or who have a positive pregnancy test result prior to receiving the first dose of IMP or RHEZ on Day 1.
* History of significant drug and/or alcohol abuse within 2 years prior to screening.
* History of or current hepatitis or carriers of HBsAg and/or anti-HCV.
* Positive urine or blood alcohol test and/or urine drug screen for substance abuse at screening (not including cannabinoids).
* History of having taken an investigational drug within 30 days preceding trial entry (ie, prior to screening).
* A history of difficulty in donating blood.
* Donation of blood or plasma within 30 days prior to dosing.
* Consumption of alcohol and/or grapefruit, grapefruit juice, Seville oranges, or Seville orange juice and related products within 72 hours prior to the first dose of IMP or RHEZ on Day 1.
* History of serious mental disorders that, in the opinion of the investigator, would exclude the subject from participating in this trial.
* Any known prior exposure to OPC-167832, delamanid or Bedaquiline.
* Participants with significant medical comorbidities that in the opinion of the investigator, should not participate in the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique R de Jager, MD, Principal Investigator — TASK Clinical Research Centre; Prof. Rodney Dawson, MD, Principal Investigator — University of Cape Town (Pty) Ltd.; Prof. Andreas Diacon, Principal Investigator — TASK Clinical Research Centre (TCRC)
Locations (3):
- South Africa (3):
  - University of Cape Town (Pty) Ltd., Cape Town, Mowbray
  - Satellite Site: Task at Brooklyn Chest Hospital, Cape Town
  - TASK Clinical Research Centre, Cape Town

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawson R, Diacon AH, De Jager V, Narunsky K, Moodley VM, Stinson KW, Liu Y, Zheng B, Hafkin J. Safety, pharmacokinetics, and early bactericidal activity of quabodepistat in combination with delamanid, bedaquiline, or both in adults with pulmonary tuberculosis: a randomised, active-controlled, open-label trial. Lancet Infect Dis. 2025 Apr;25(4):435-444. doi: 10.1016/S1473-3099(24)00601-7. Epub 2024 Nov 26. PMID 39612928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at two investigative sites in South Africa from 18 October 2018 to 11 March 2022.
Pre-assignment Details: Participants with uncomplicated, smear-positive, drug-susceptible pulmonary tuberculosis were enrolled in two stages. Stage 1: A total of 76 participants were randomized in 4 cohorts to receive either OPC-167832 10 milligrams (mg), 30 mg, 90 mg & 3 mg or a combination of rifampicin, isoniazid, ethambutol, and pyrazinamide (RHEZ). Stage 2: A total of 46 participants were randomized in 4 groups to receive OPC-167832+delamanid, OPC-167832+bedaquilline (BDQ), OPC-167832+delamanid+BDQ or RHEZ.
Groups:
- Stage 1: 10 mg OPC-167832: Participants received OPC-167832, 10 milligrams (mg), orally, once daily (QD), from Day 1 through Day 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
- Stage 1: RHEZ: Participants received a single dose of RHEZ (each tablet containing 150 mg rifampicin, 75 mg isoniazid, 400 mg pyrazinamide, and 275 mg ethambutol), orally, QD from Day 1 through Day 20.
- Stage 2: 30 mg OPC-167832 + 400 mg BDQ: Participants received OPC-167832, 30 mg, in combination with BDQ, orally, QD, from Day 1 through Day 14. Participants received a loading dose of 700 mg BDQ on Day 1 and 500 mg on Day 2. BDQ was then administered at a dose of 400 mg, QD, orally from Days 3 to 14. After Day 14, participants received RHEZ according to the local standard of care regimen up to Day 20.
Period: Overall Study
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ | Stage 2: RHEZ
Started | 14 | 14 | 17 | 14 | 17 | 14 | 14 | 14 | 4
Efficacy Analysis Set/ MITT Set (Modified Intent-to-Treat (MITT) Analysis Set included randomized participants who were agar media culture positive at baseline (either at Day -2 or at Day -1, or both), received any dose of investigational medicinal product (IMP), and had at least one post-baseline colony forming unit (CFU) count value.) | 14 | 11 | 14 | 14 | 15 | 11 | 11 | 12 | 4
Safety Analysis Set (Safety Analysis Set included participants who were randomized and took any dose of IMP.) | 14 | 14 | 17 | 14 | 16 | 13 | 13 | 14 | 4
Pharmacokinetic (PK) Analysis Set (PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration.) | 14 | 14 | 17 | 14 | 11 | 13 | 13 | 14 | 4
Completed | 14 | 14 | 14 | 13 | 16 | 10 | 9 | 11 | 4
Not Completed | 0 | 0 | 3 | 1 | 1 | 4 | 5 | 3 | 0
Not completed — Reason not Specified | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non-Covid Related Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Covid Related Adverse Event | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set included participants who were randomized into the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ | Stage 2: RHEZ | Total
Number analyzed (Participants) | 14 | 14 | 17 | 14 | 17 | 14 | 14 | 14 | 4 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (14.6) | 34.9 (12.8) | 36.2 (13.3) | 37.2 (15.6) | 33.4 (10.9) | 34.1 (9.9) | 29.8 (8.9) | 30.1 (8.2) | 31.3 (9.5) | 33.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 8 | 4 | 5 | 2 | 2 | 4 | 1 | 38
  Male | 10 | 6 | 9 | 10 | 12 | 12 | 12 | 10 | 3 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 12 | 17 | 14 | 15 | 14 | 14 | 14 | 4 | 118
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 7 | 11 | 6 | 8 | 7 | 10 | 9 | 3 | 69
  Other | 6 | 7 | 5 | 8 | 9 | 7 | 4 | 5 | 1 | 52
  White | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Change From Baseline in TB Bacterial Load in Sputum as a Measure of Early Bactericidal Activity (EBA)
Description: Bacterial load in sputum at each collection time point was measured by CFU counts on agar media culture. EBA was determined by the rate of decline per day in log10CFU/mL during the first 14 days of treatment. Change from baseline in log 10 CFU was calculated as post-baseline minus baseline. A larger EBA in positive direction indicates a better drug effect.
Time Frame: Baseline to Day 14
Population: MITT Analysis Set included randomized participants who were agar media culture positive at baseline (either at Day -2 or at Day -1, or both), received any dose of IMP, and had at least one post-baseline CFU count value. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: sputum log10CFU/mL
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ
Number analyzed (Participants) | 14 | 10 | 13 | 11 | 14
sputum log10CFU/mL | -1.93 (0.98) | -2.12 (1.01) | -2.08 (0.75) | -1.69 (1.15) | -2.79 (0.96)
Statistical Analysis 1: Comparison: Stage 1: 10 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.689, 95% CI 2-sided [0.485 to 0.939] — The confidence interval for the EBA ratio is estimated using Fieller's method
Statistical Analysis 2: Comparison: Stage 1: 10 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.689, 95% CI 2-sided [0.467 to 0.911] — The confidence interval for the EBA ratio is estimated using Taylor's method
Statistical Analysis 3: Comparison: Stage 1: 30 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.759, 95% CI 2-sided [0.517 to 1.051] — The confidence interval for the EBA ratio is estimated using Fieller's method
Statistical Analysis 4: Comparison: Stage 1: 30 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.759, 95% CI 2-sided [0.497 to 1.020] — The confidence interval for the EBA ratio is estimated using Taylor's method
Statistical Analysis 5: Comparison: Stage 1: 90 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.745, 95% CI 2-sided [0.567 to 0.973] — The confidence interval for the EBA ratio is estimated using Fieller's method
Statistical Analysis 6: Comparison: Stage 1: 90 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.745, 95% CI 2-sided [0.547 to 0.943] — The confidence interval for the EBA ratio is estimated using Taylor's method
Statistical Analysis 7: Comparison: Stage 1: 3 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.605, 95% CI 2-sided [0.353 to 0.896] — The confidence interval for the EBA ratio is estimated using Fieller's method
Statistical Analysis 8: Comparison: Stage 1: 3 mg OPC-167832 vs Stage 1: RHEZ; Test type: Superiority; EBA Ratio = 0.605, 95% CI 2-sided [0.338 to 0.871] — The confidence interval for the EBA ratio is estimated using Taylor's method

2. Primary Outcome: Stage 1 and Stage 2: Maximum (Peak) Plasma Concentration (Cmax) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 14 | 14 | 14 | 17 | 13 | 13 | 14
nanogram per milliliter (ng/mL) | 20.7 (6.92) | 53.7 (9.16) | 128 (50.5) | 391 (116) | 157 (44.1) | 154 (39.6) | 140 (41.2)

3. Primary Outcome: Stage 1 and Stage 2: Cmax at Steady-state (Cmax,ss) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
ng/mL | 28.2 (10.9) | 67.3 (11.9) | 190 (63.6) | 492 (99.8) | 208 (60.5) | 175 (31.3) | 183 (51.9)

4. Primary Outcome: Stage 1 and Stage 2: Time to Cmax (Tmax) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 14 | 14 | 14 | 17 | 13 | 13 | 14
hours | 3.17 [2.17 to 4.17] | 4.15 [1.17 to 5.15] | 3.15 [2.15 to 5.17] | 3.25 [2.13 to 5.17] | 2.83 [1.83 to 4.83] | 3.17 [1.17 to 5.18] | 3.83 [1.80 to 7.90]

5. Primary Outcome: Stage 1 and Stage 2: Tmax of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
hours | 3.17 [1.18 to 5.17] | 3.15 [1.15 to 5.13] | 3.13 [2.13 to 5.13] | 3.17 [2.13 to 5.13] | 2.83 [1.82 to 5.83] | 3.13 [2.17 to 4.25] | 2.83 [1.83 to 4.85]

6. Primary Outcome: Stage 1 and Stage 2: Area Under the Concentration-Time Curve (AUC) From Time Zero to Time t (the Last Observable Concentration, Here t=24) (AUC0-24), for OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram.hour per milliliter (ng*h/mL)
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 14 | 13 | 14 | 17 | 12 | 13 | 14
nanogram.hour per milliliter (ng*h/mL) | 178 (65.1) | 569 (102) | 1290 (532) | 4050 (1240) | 1450 (392) | 1490 (490) | 1420 (378)

7. Primary Outcome: Stage 1 and Stage 2: AUC Calculated Over the Dosing Interval at Steady-state (AUCτ) for OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
ng*h/mL | 349 (143) | 874 (127) | 2490 (928) | 5690 (1010) | 2500 (709) | 2020 (563) | 2000 (730)

8. Primary Outcome: Stage 1 and Stage 2: Terminal-phase Elimination Half-life (t1/2,z) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Description: T1/2,z is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose. Half-life (T1/2) is determined in the terminal phase after drug administration, which is calculated from the relationship T1/2 = ln2/λz where λz is the terminal-phase slope obtainable from non-compartmental analysis (NCA). The values reported for this outcome measure (OM) are estimates and not actual observed data.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 9 | 10 | 10
hours | 22.3 [10.3 to 36.7] | 15.3 [9.2 to 22.5] | 14.2 [5.6 to 29.1] | 14.4 [9.8 to 30.1] | 14.4 [13.3 to 20.4] | 14.7 [6.2 to 22.1] | 11.2 [6.8 to 19.1]

9. Primary Outcome: Stage 1 and Stage 2: Apparent Clearance From Plasma at Steady-state (CLss/F) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/minute (min)
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
mL/minute (min) | 164 (62.6) | 195 (28.8) | 231 (91.8) | 272 (53.8) | 215 (61.0) | 269 (88.5) | 283 (103)

10. Primary Outcome: Stage 1 and Stage 2: Accumulation Ratio of Cmax (RCmax) for OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
ratio | 1.39 (0.381) | 1.26 (0.167) | 1.56 (0.399) | 1.36 (0.362) | 1.34 (0.349) | 1.23 (0.191) | 1.30 (0.244)

11. Primary Outcome: Stage 1 and Stage 2: Accumulation Ratio of AUC (RAUC) for OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 13 | 14 | 14 | 11 | 10 | 11
ratio | 1.99 (0.550) | 1.60 (0.289) | 2.01 (0.565) | 1.55 (0.416) | 1.70 (0.378) | 1.47 (0.314) | 1.36 (0.237)

12. Primary Outcome: Stage 1 and Stage 2: Cmax Normalized to Dose (Cmax/Dose) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (ng/mL)/mg
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
(ng/mL)/mg | 9.42 (3.63) | 6.73 (1.19) | 6.34 (2.12) | 5.46 (1.11) | 6.94 (2.02) | 5.85 (1.04) | 6.10 (1.73)

13. Primary Outcome: Stage 2: AUCτ Normalized to Dose (AUCτ/Dose) of OPC-167832 When Administered Alone (Stage 1) and in Combination With Delamanid, and BDQ (Stage 2)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (ng*h/mL)/mg
Arm/Group | Stage 1: 3 mg OPC-167832 | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 11 | 10 | 11
(ng*h/mL)/mg | 116 (47.6) | 87.4 (12.7) | 82.8 (30.9) | 63.3 (11.2) | 83.5 (23.6) | 67.2 (18.8) | 66.5 (24.3)

14. Primary Outcome: Stage 2: Cmax of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14
ng/mL | 181 (41.8) | 198 (57.5)

15. Primary Outcome: Stage 2: Cmax,ss of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
ng/mL | 401 (102) | 442 (188)

16. Primary Outcome: Stage 2: Tmax of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14
hours | 3.82 [1.83 to 5.83] | 4.82 [2.83 to 7.90]

17. Primary Outcome: Stage 2: Tmax of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
hours | 3.83 [1.83 to 5.83] | 3.83 [2.70 to 7.83]

18. Primary Outcome: Stage 2: AUC0-24 of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 12 | 14
ng.h/mL | 2140 (613) | 2440 (957)

19. Primary Outcome: Stage 2: AUCτ of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
ng*h/mL | 5460 (1620) | 5860 (2310)

20. Primary Outcome: Stage 2: T1/2,z of Delamanid
Description: T1/2,z is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose. Half-life (T1/2) is determined in the terminal phase after drug administration, which is calculated from the relationship T1/2 = ln2/λz where λz is the terminal-phase slope obtainable using the NCA method. The values reported for this OM are estimates and not actual observed data.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 9 | 9
hours | 25.4 [16.3 to 38.4] | 25.1 [17.6 to 56.4]

21. Primary Outcome: Stage 2: CLss/F of Delamanid From Plasma
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
mL/min | 983 (264) | 966 (330)

22. Primary Outcome: Stage 2: RCmax of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
ratio | 2.26 (0.647) | 2.19 (0.601)

23. Primary Outcome: Stage 2: RAUC of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
ratio | 2.69 (0.683) | 2.49 (0.897)

24. Primary Outcome: Stage 2: Cmax/Dose of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (ng/mL)/mg
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
(ng/mL)/mg | 1.34 (0.339) | 1.47 (0.625)

25. Primary Outcome: Stage 2: AUCτ/Dose of Delamanid
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (ng*h/mL)/mg
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
(ng*h/mL)/mg | 18.2 (5.40) | 19.5 (7.71)

26. Primary Outcome: Stage 2: Cmax of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 12 | 14
ng/mL | 5150 (1860) | 5750 (2320)

27. Primary Outcome: Stage 2: Cmax,ss of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
ng/mL | 5030 (1850) | 6080 (1660)

28. Primary Outcome: Stage 2: Tmax of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 12 | 14
hours | 5.17 [4.13 to 8.15] | 4.83 [3.82 to 7.90]

29. Primary Outcome: Stage 2: Tmax of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
hours | 5.17 [3.15 to 5.20] | 4.85 [4.83 to 5.82]

30. Primary Outcome: Stage 2: AUC0-24 of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 12 | 13
ng*h/mL | 44900 (12800) | 47000 (15600)

31. Primary Outcome: Stage 2: AUCτ of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
ng*h/mL | 55900 (16000) | 66000 (19200)

32. Primary Outcome: Stage 2: T1/2,z of Bedaquiline
Description: T1/2,z is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose. Half-life (T1/2) is determined in the terminal phase after drug administration, which is calculated from the relationship T1/2 = ln2/λz where λz is the terminal-phase slope obtainable using the NCA method. The values reported for this OM are estimates and not actual observed data. Hence, the value might not lie within the sampling timepoints provided in the timeframe.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 5 | 7
hours | NA [14.4 to 139.7] — For the parameter that was not reported, due to less than 50% of the subjects having enough data to estimate the parameter, the descriptive statistic was not determined and not reported. | 81.1 [54.2 to 155.4]

33. Primary Outcome: Stage 2: CLss/F of BDQ From Plasma
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
mL/min | 140 (85.9) | 109 (31.4)

34. Primary Outcome: Stage 2: Cmax/Dose of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (ng/mL)/mg
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
(ng/mL)/mg | 12.6 (4.62) | 15.2 (4.14)

35. Primary Outcome: Stage 2: AUCτ/Dose of Bedaquiline
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: (ng*h/mL)/mg
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
(ng*h/mL)/mg | 140 (40.0) | 165 (48.0)

36. Primary Outcome: Stage 1 and Stage 2: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs were all AEs which started after the start of randomized study drug treatment or if the event was continuous from baseline and was serious, study drug-related, or resulted in death, discontinuation, interruption, or reduction of study therapy.
Time Frame: From first dose of study drug to end of follow up period (up to 34 days)
Population: Safety Analysis Set included participants who were randomized and received any dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ | Stage 2: RHEZ
Number analyzed (Participants) | 14 | 14 | 17 | 14 | 16 | 13 | 13 | 14 | 4
Participants | 10 | 13 | 13 | 11 | 15 | 9 | 11 | 9 | 3

37. Primary Outcome: Stage 1 and Stage 2: Number of Participants With Clinically Significant Changes in Vital Sign Values
Time Frame: From first dose of study drug to end of follow up period (up to 34 days)
Population: Safety Analysis Set included participants who were randomized and received any dose of IMP. Number analyzed is the number of participants with data available for analysis for each specified vital sign parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ | Stage 2: RHEZ
Number analyzed (Participants) | 14 | 14 | 17 | 14 | 16 | 13 | 13 | 14 | 4
Participants
  Heart Rate: > 120 beats per minute (bpm) and >= 15 bpm Change from Baseline | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Diastolic Blood Pressure: < 50 mmHg and >= 15 mmHg Decrease from Baseline | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0
  Systolic Blood Pressure: < 90 mmHg and >= 20 mmHg Decrease from Baseline | 1 | 3 | 2 | 2 | 0 | 1 | 1 | 1 | 0
  Weight: >= 5% Increase from Baseline: number analyzed (Participants) | 14 | 14 | 16 | 13 | 16 | 13 | 13 | 14 | 4
  Weight: >= 5% Increase from Baseline | 3 | 4 | 2 | 1 | 9 | 0 | 5 | 2 | 2

38. Primary Outcome: Stage 1 and Stage 2: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Time Frame: From first dose of study drug to end of follow up period (up to 34 days)
Population: Safety Analysis Set included participants who were randomized and received any dose of IMP. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ | Stage 2: RHEZ
Number analyzed (Participants) | 14 | 14 | 14 | 13 | 16 | 11 | 11 | 12 | 4
Participants
  Rhythm: Ventricular Premature Beat | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  ST/T Morphology: Myocardial Ischemia | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ST/T Morphology: Symmetrical T-wave Inversion | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

39. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in Lipoarabinomannan (LAM) in the Mycobacteria Growth Indicator Tube® (MGIT) System
Description: LAM is a key component of the M. tuberculosis cell wall and the decline of sputum LAM concentrations has been shown to correlate closely with CFU decreases in sputum counted on agar media during the first 14 days of TB treatment. Sputum LAM concentration at each collection time point was measured using MGIT system. Baseline LAM was calculated as the log 10 of the average from Day -2 and Day -1 and the change from baseline in log10 was calculated as post-baseline minus baseline for each parameter.
Time Frame: Baseline to Day 14
Population: MITT Analysis Set included randomized participants who were agar media culture positive at baseline (either at Day -2 or at Day -1, or both), received any dose of IMP, and had at least one post-baseline CFU count value. Overall number of participants analyzed is the number of participants with data available for analysis. As pre-specified in the protocol and SAP, for Stage 2 data for participants in RHEZ arm was not included in this analysis.
Measure: Mean (Standard Deviation); unit: log10 LAM picograms (pg)/ml
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 14 | 11 | 14 | 13 | 15 | 11 | 10 | 10
log10 LAM picograms (pg)/ml
  Raw | -1.52 (0.79) | -1.41 (0.75) | -1.44 (0.67) | -1.35 (0.76) | -1.19 (0.75) | -1.93 (1.22) | -0.97 (0.62) | -2.06 (1.03)
  Processed | -1.43 (1.07) | -1.55 (0.90) | -1.40 (0.77) | -1.42 (0.74) | -1.05 (0.61) | -2.05 (1.26) | -0.87 (0.66) | -1.84 (1.39)

40. Secondary Outcome: Stage 1 and Stage 2: Change From Baseline in Time to Detection (TTD) in the MGIT System
Description: TTD is the time from start of inoculation of a sputum sample until a MGIT machine detects a positive signal during the 42-day incubation period. One TTD measurement, reported in days and hours was taken at each of the visits at Days -2, -1, 2, 4, 6, 8, 10, 12 and 14. TTD values were then calculated as "days + hours/24" to be used in deriving the analysis values of TTD. Each sample collected from Day -2 to Day 14 were inoculated for 42 days. Baseline TTD was derived using Day -2 and Day -1 MGIT culture with a pure positive result for Mycobacterium tuberculosis. Postbaseline TTD analysis values from Day 1 were derived based on the MGIT culture result as follows: If MGIT culture result was negative for MTB complex, TTD was set to 42 days; If the MGIT culture was pure positive for MTB, but the TTD took longer than 42 days, TTD was capped at 42 days.
Time Frame: Day 1 to Day 14 of treatment period + 42 days of inoculation period (up to 56 days)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 14 | 11 | 13 | 13 | 15 | 11 | 10 | 10
days | 4.28 (2.88) | 9.54 (13.63) | 18.15 (15.06) | 3.33 (2.74) | 7.44 (1.65) | 8.93 (10.31) | 5.33 (2.54) | 14.26 (13.57)

41. Secondary Outcome: Stage 2: Change From Baseline in TB Bacterial Load in Sputum as a Measure of EBA
Description: as for outcome 1
Time Frame: Baseline to Day 14
Population: MITT Analysis Set included randomized participants who were agar media culture positive at baseline (either at Day -2 or at Day -1, or both), received any dose of IMP, and had at least one post-baseline CFU count value. Overall number analyzed is the number of participants with data available for analysis. As pre-specified in the protocol and SAP, for Stage 2 data for participants in RHEZ arm was not included in this analysis.
Measure: Mean (Standard Error); unit: Sputum log10 CFU/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 8 | 9 | 7
Sputum log10 CFU/mL | -2.17 (1.83) | -1.97 (1.29) | -2.73 (1.51)
Statistical Analysis 1: Comparison: Stage 2: 30 mg OPC-167832 + 300 mg Delamanid vs Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ; Test type: Superiority; EBA Ratio = 1.256, 95% CI 2-sided [0.626 to 3.175] — The confidence interval for the EBA ratio is estimated using Fieller's method
Statistical Analysis 2: Comparison: Stage 2: 30 mg OPC-167832 + 300 mg Delamanid vs Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ; Test type: Superiority; EBA Ratio = 1.256, 95% CI 2-sided [0.362 to 2.151] — The confidence interval for the EBA ratio is estimated using Taylor's method
Statistical Analysis 3: Comparison: Stage 2: 30 mg OPC-167832 + 400 mg BDQ vs Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ; Test type: Superiority; EBA Ratio = 1.385, 95% CI 2-sided [0.736 to 2.656] — The confidence interval for the EBA ratio is estimated using Fieller's method
Statistical Analysis 4: Comparison: Stage 2: 30 mg OPC-167832 + 400 mg BDQ vs Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ; Test type: Superiority; EBA Ratio = 1.385, 95% CI 2-sided [0.564 to 2.206] — The confidence interval for the EBA ratio is estimated using Taylor's method

42. Secondary Outcome: Stage 2: Plasma Concentration of Rifampin
Time Frame: 2 hours and 6 hours post-dose on Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: RHEZ
Number analyzed (Participants) | 4
ng/mL
  2 hours Post-dose | 4020 (2450)
  6 hours Post-dose | 1880 (811)

43. Secondary Outcome: Stage 1: Plasma Concentration of Isoniazid
Time Frame: 2 hours and 6 hours post-dose on Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per millilitre (ug/mL)
Arm/Group | Stage 1: RHEZ
Number analyzed (Participants) | 11
microgram per millilitre (ug/mL)
  2 hours Post-dose | 4.16 (1.45)
  6 hours Post-dose | 1.58 (0.837)

44. Secondary Outcome: Stage 2: Cmax of DM-6705
Description: DM-6705 is a metabolite of delamanid.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14
ng/mL | 10.3 (10.5) | 14.6 (11.6)

45. Secondary Outcome: Stage 2: Cmax,ss of DM-6705
Description: DM-6705 is a metabolite of delamanid.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11
ng/mL | 84.0 (27.5) | 112 (51.9)

46. Secondary Outcome: Stage 2: Tmax of DM-6705
Description: DM-6705 is a metabolite of delamanid.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1; Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 14
hours
  Day 1 | 4.82 [1.83 to 23.63] | 4.83 [1.83 to 23.58]
  Day 14: number analyzed (Participants) | 11 | 11
  Day 14 | 4.83 [0.33 to 7.83] | 4.85 [2.70 to 11.85]

47. Secondary Outcome: Stage 2: AUC0-24 for DM-6705
Description: DM-6705 is a metabolite of delamanid.
Time Frame: as for outcome 46
Population: PK Analysis Set included all participants who received at least one dose of IMP and had 1 quantifiable drug concentration. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 12 | 14
ng*h/mL
  Day 1 | 103 (54.2) | 166 (124)
  Day 14: number analyzed (Participants) | 11 | 11
  Day 14 | 1620 (458) | 1980 (850)

48. Secondary Outcome: Stage 2: T1/2,z of DM-6705
Description: T1/2,z is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose. Half-life (T1/2) was determined in the terminal phase after drug administration, which was calculated from the relationship T1/2 = ln2/λz where λz is the terminal-phase slope obtainable using the NCA method. The values reported for this OM are estimates and not actual observed data. Hence, the value might not lie within the sampling timepoints provided in the timeframe.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 5 | 4
hours | NA [90.2 to 509.1] — For the parameter that was not reported, due to less than 50% of the subjects having enough data to estimate the parameter, the descriptive statistic was not determined and not reported. | NA [95.8 to 1219.9] — For the parameter that was not reported, due to less than 50% of the subjects having enough data to estimate the parameter, the descriptive statistic was not determined and not reported.

49. Secondary Outcome: Stage 2: Cmax of N-Desmethyl Bedaquiline
Description: N-Desmethyl Bedaquiline is a metabolite of BDQ.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours postdose on Day 1
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 12
ng/mL | 95.4 (44.7) | 88.2 (17.5)

50. Secondary Outcome: Stage 2: Cmax,ss of N-Desmethyl Bedaquiline
Description: N-Desmethyl Bedaquiline is a metabolite of BDQ.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
ng/mL | 489 (154) | 575 (112)

51. Secondary Outcome: Stage 2: Tmax of N-Desmethyl Bedaquiline
Description: N-Desmethyl Bedaquiline is a metabolite of BDQ.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours (±15 minutes) postdose on Day 1; Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
hours
  Day 1 | 23.93 [6.17 to 24.05] | 11.86 [7.82 to 23.88]
  Day 14 | 15.08 [0.00 to 48.0] | 7.83 [3.83 to 23.63]

52. Secondary Outcome: Stage 2: AUC0-24 for N-Desmethyl Bedaquiline
Description: N-Desmethyl Bedaquiline is a metabolite of BDQ.
Time Frame: as for outcome 46
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 10 | 11
ng*h/mL
  Day 1 | 1380 (731) | 1410 (326)
  Day 14 | 10100 (3080) | 11800 (1920)

53. Secondary Outcome: Stage 2: Number of Participants With TEAEs on Administration of OPC-167832 in Combination With Delamanid and/or Bedaquiline
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. TEAEs were all adverse events which started after the start of randomized study drug treatment or if the event was continuous from baseline and was serious, study drug-related, or resulted in death, discontinuation, interruption, or reduction of study therapy.
Time Frame: From first dose of study drug to end of follow up period (up to 34 days)
Population: Safety Analysis Set included participants who were randomized and received any dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 13 | 14
Participants | 9 | 11 | 9

54. Secondary Outcome: Stage 2: Number of Participants With Clinically Significant Vital Sign Changes on Administration of OPC-167832 in Combination With Delamanid and/or Bedaquiline
Time Frame: From first dose of study drug to end of follow up period (up to 34 days)
Population: Safety Analysis Set included participants who were randomized and received any dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 13 | 13 | 14
Participants
  Heart Rate: > 120 bpm and >= 15 bpm change from baseline | 0 | 1 | 0
  Diastolic blood pressure: < 50 mmHg and >= 15 mmHg decrease from baseline | 0 | 2 | 0
  Systolic blood pressure: < 90 mmHg and >= 20 mmHg decrease from baseline | 1 | 1 | 1
  Weight: >= 5% increase from baseline | 0 | 5 | 2

55. Secondary Outcome: Stage 2: Number of Participants With Clinically Significant Changes in ECG Evaluations on Administration of OPC-167832 in Combination With Delamanid and/or Bedaquiline
Time Frame: From first dose of study drug to end of follow up period (up to 34 days)
Population: Safety Analysis Set included participants who were randomized and received any dose of IMP. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ
Number analyzed (Participants) | 11 | 11 | 12
Participants
  Rhythm: Ventricular Premature Beat | 0 | 0 | 0
  ST/T Morphology: Myocardial Ischemia | 0 | 0 | 0
  ST/T Morphology: Symmetrical T-wave Inversion | 0 | 0 | 0

56. Other Pre Specified Outcome: Correlation of QT Interval and Plasma Concentrations of OPC-167832 and/or Delamanid and/or Bedaquiline
Time Frame: Day 1 and Day 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of follow up period (up to approximately 34 days in each Stage 1 and Stage 2)
Description: Safety Analysis Set included participants who were randomized and received any dose of IMP.
Arm/Group | Stage 1: 10 mg OPC-167832 | Stage 1: 30 mg OPC-167832 | Stage 1: 90 mg OPC-167832 | Stage 1: 3 mg OPC-167832 | Stage 1: RHEZ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid | Stage 2: 30 mg OPC-167832 + 400 mg BDQ | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ | Stage 2: RHEZ
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/17 | 0/14 | 0/16 | 0/13 | 0/13 | 0/14 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/17 | 1/14 | 0/16 | 0/13 | 2/13 | 0/14 | 0/4
Other Adverse Events (participants affected / at risk) | 10/14 | 13/14 | 13/17 | 10/14 | 15/16 | 9/13 | 11/13 | 9/14 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: 10 mg OPC-167832 (N=14) | Stage 1: 30 mg OPC-167832 (N=14) | Stage 1: 90 mg OPC-167832 (N=17) | Stage 1: 3 mg OPC-167832 (N=14) | Stage 1: RHEZ (N=16) | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid (N=13) | Stage 2: 30 mg OPC-167832 + 400 mg BDQ (N=13) | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ (N=14) | Stage 2: RHEZ (N=4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: 10 mg OPC-167832 (N=14) | Stage 1: 30 mg OPC-167832 (N=14) | Stage 1: 90 mg OPC-167832 (N=17) | Stage 1: 3 mg OPC-167832 (N=14) | Stage 1: RHEZ (N=16) | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid (N=13) | Stage 2: 30 mg OPC-167832 + 400 mg BDQ (N=13) | Stage 2: 30 mg OPC-167832 + 300 mg Delamanid + 400 mg BDQ (N=14) | Stage 2: RHEZ (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival Irritation (Eye disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 3 | 0
Catheter Site Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Injection Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel Puncture Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea Capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver Function Test Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 0
Headache (Nervous system disorders) | 3 | 4 | 2 | 3 | 2 | 2 | 4 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 3 | 2 | 6 | 0 | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Contractions Involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03678688/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03678688/SAP_001.pdf